CLINICAL TRIAL: NCT04238078
Title: Investigation of Taste Function and Eating Habits in Women With Polycystic Ovary Syndrome
Brief Title: Taste Function and Eating Habits in Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Okan Bulent Yildiz, Professor of Medicine, Hacettepe University
Other Study IDs: 17697
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Contraceptive Agents; Contraceptives, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polycystic ovary syndrome: Women with PCOS diagnosed according to Rotterdam criteria
  Interventions: Drug: Contraceptive
- Healthy control: Healthy women without any feature of ovulatory dysfunction or androgen excess

INTERVENTIONS:
Drug: Contraceptive — Oral contraceptive pill
  Other Names: birth control pill
  Groups: Polycystic ovary syndrome

SUMMARY:
This study evaluates taste function and eating habits in patients with PCOS compared to healthy women and before and after oral contraceptive use.

DETAILED DESCRIPTION:
The objective of this study is to investigate the taste function and eating habits in patients with PCOS in comparison with healthy women at baseline and after routine use of an oral contraceptive (2mg ethinylestradiol and 0.03mg dienogest) along with general lifestyle advice for three months.

Patients with diagnosis of PCOS (Rotterdam criteria) will be recruited from Hacettepe University outpatient clinics. Along with clinical, hormonal and biochemical evaluation, taste function and eating habit tests will be performed at baseline both in patients and healthy volunteers. These tests will be repeated in women with PCOS after 3 months of oral contraceptive use.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS (Rotterdam criteria) who will receive oral contraceptive pill for long-term management

Exclusion Criteria:

* Any systemic illness
* Any other medication use
* Age<18 or >35 years
* Pregnant or nursing
* Untreated hypothyroidism or hyperthyroidism
* Known rhinoplasty or nasal surgery
* Known defect in smell or taste function
* Being active smoker.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with PCOS
Study Population: Outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Taste function | Three months
  Taste function assessed by use of taste strip test

SECONDARY OUTCOMES:
Eating habits | Three months
  Eating habits assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Yildiz, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data generated during the study will be available from the principal investigator on reasonable request

REFERENCES:
- [Result] Simchen U, Koebnick C, Hoyer S, Issanchou S, Zunft HJ. Odour and taste sensitivity is associated with body weight and extent of misreporting of body weight. Eur J Clin Nutr. 2006 Jun;60(6):698-705. doi: 10.1038/sj.ejcn.1602371. Epub 2006 Jan 25. PMID 16435003
- [Result] Wolf A, Varga L, Wittibschlager L, Renner B, Mueller CA. A self-administered test of taste function using "Taste Strips". Int Forum Allergy Rhinol. 2016 Apr;6(4):362-6. doi: 10.1002/alr.21681. Epub 2015 Dec 3. PMID 26633243